CLINICAL TRIAL: NCT02949635
Title: Risks of Death, Hospital Readmission, and Institutionalization After Hospitalization in Acute Geriatric Unit
Brief Title: Patient Outcomes After Hospitalization in Acute Geriatric Unit
Acronym: DAMAGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014_23; 2014-A01670-47 (Other: ID-RCB number, ANSM); API 13-19-002 (Other: PHRC number, DGOS)
Record Dates: First submitted 2016-08-23; First posted 2016-10-31 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Geriatric Disorder
Keywords: Aged; Patient readmission; Geriatric Assessment; Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Three events can be considered of major importance for patients after a hospitalization in an AGU: death, hospital readmission, and institutionalization. Current published data do not allow the clinician to simultaneously estimate the risk of hospital readmission, institutionalization and death of an older patient according to his/her characteristics and various complications that occurred during the hospitalization. However, clinicians often need to estimate these risks at hospital discharge to adapt their therapeutic choices, their proposals post-hospital care, and provide reliable and fair information to the patient and his relatives.

Estimating simultaneously the hazard for each of these three events can be complex. Indeed, a death event hinder the observation of re-hospitalization or institutionalization if death occurs before these events. The death should be considered a competing risk in these analyzes. Hospital readmission may modify the risk of death or institutionalization and should be considered as an intermediate factor for these event. This complexity cannot be accounted with classical statistical models, like logistic regression models.

The purpose of this study is to use more appropriate statistical models (multi-state models) to better estimate simultaneously the risks of hospital readmission, institutionalization, and death of a patient given after hospitalization in AGU, and to show that accuracy of these estimations can be improved by taking into account complications that occurred during the stay in AGU.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years and over
* Hospitalized in Acute Geriatric Unit
* Covered by a health insurance

Exclusion Criteria:

* Refusal to participate to the study, as expressed by the patient or his/her next of kin

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All consecutive incident patients aged 75 years and older hospitalized in an acute geriatric unit will be eligible and included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3532 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of death after discharge | 3 months

SECONDARY OUTCOMES:
Number of death after discharge | 12 months
Number of rehospitalization after discharge | at 3 and 12 months
Number of institutionalization (NH admissions) | at 12 months
Number of nosocomial infectious diseases during the index hospitalization | 60 days
Duration of clostridium difficile infection | 60 days
Length of stay of the index hospitalization | 60 days
  The exact duration for this outcome will correspond to the duration of the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Beuscart, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (6):
- France (6):
  - CHU d'Amiens, Amiens
  - CH Beauvais, Beauvais
  - CHU Caen, Caen
  - Hôpital Cardiologique, CHRU, Lille
  - GHICL, Saint Philibert, Lomme
  - CH Saint Quentin, Saint-Quentin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prod'homme C, Deschasse G, Visade F, Hennion C, Charpentier A, Gaxatte C, Bloch F, Delecluse C, Puisieux F, Beuscart JB. Palliative use of midazolam in acute geriatric units: a multicenter ambispective study. BMC Geriatr. 2025 Apr 10;25(1):241. doi: 10.1186/s12877-025-05860-6. PMID 40211151
- [Derived] Deschasse G, Charpentier A, Prod'homme C, Genin M, Delecluse C, Gaxatte C, Gerard C, Bukor Z, Devulder P, Couvreur LA, Bloch F, Puisieux F, Visade F, Beuscart JB. Transition to Comfort Care Only and End-of-Life Trajectories in an Acute Geriatric Unit: A Secondary Analysis of the DAMAGE Cohort. J Am Med Dir Assoc. 2022 Sep;23(9):1492-1498. doi: 10.1016/j.jamda.2022.04.016. Epub 2022 May 21. PMID 35609637
- [Derived] Deschasse G, Bloch F, Drumez E, Charpentier A, Visade F, Delecluse C, Loggia G, Lescure P, Attier-Zmudka J, Bloch J, Gaxatte C, Van Den Berghe W, Puisieux F, Beuscart JB. Development of a Predictive Score for Mortality at 3 and 12 Months After Discharge From an Acute Geriatric Unit as a Trigger for Advanced Care Planning. J Gerontol A Biol Sci Med Sci. 2022 Aug 12;77(8):1665-1672. doi: 10.1093/gerona/glab217. PMID 34375411